CLINICAL TRIAL: NCT02810938
Title: Prospective Atrial Flutter Ablation Registry Investigating IntellaTip Mifi XP 8 mm Technology and Maximum Voltage-guided (MVG) Isthmus Ablation Approach
Brief Title: MIFI Flutter Registry - Ablation of Atrial Flutter With IntellaTip Sensor Technology
Acronym: MIFI
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MIFI
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Atrial Flutter
Keywords: Ablation; Mifi technology; maximum voltage-guided ablation
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ablation of atrial flutter — Ablation of atrial flutter using IntellaTip Mifi 8 mm technology in combination with Maximum voltage-guided ablation approach
  Other Names: Isthmus ablation

SUMMARY:
* Prospective Atrial Flutter Ablation Registry investigating IntellaTip Mifi XP 8 mm technology and MVG isthmus ablation approach
* Design: National, multi-centre, prospective observational registry documenting right atrial isthmus ablation
* Observational treatment: Combination of MVG ablation strategy and the IntellaTip Mifi XP 8 mm sensor technology
* Duration: Patients will be followed for 6 months post-ablation

DETAILED DESCRIPTION:
The MIFI Flutter Registry is a non-interventional, multi-centre, prospective registry in consecutive patients with atrial flutter and indication for right atrial isthmus ablation. The registry is an observational study and patient's participation in this study has no impact on his/her indication for treatment, diagnostics or therapy. Patients are supposed to be treated according to current guidelines and the site's internal directives.

Treatment pattern and treatment initiation, continuation or changes are solely at the discre-tion of the physician and the patient. There will be no attempt to influence the treatment patterns of any individual treating physician. All drug prescriptions will be in the usual standard of care. Participation in the registry will in no way influence payment or reimbursement for any treatment received by subjects during the study.

A minimum of 10 hospitals in Germany treating atrial flutter and using the Maximum voltage-guided (MVG) ablation technique are eligible for participation. The enrolment period is estimated to be 6 months.

Eligible are all patients with atrial flutter, who will visit consecutively a participating site of the MIFI Flutter Registry. It is planned to enrol approximately 120 patients in total.

The follow-ups of patients will be performed using a standardized patient interview (telephone call) at 6 months by Institut für Herzinfarktforschung (IHF). In case of relevant complications, the treating physician is asked to provide medical records for verification. If the patient is not accessible by phone, local registration offices will be contacted for further information.

ELIGIBILITY:
Inclusion Criteria:

* Atrial flutter and clinical indication for atrial flutter (AFL) ablation
* 18+ years
* Written informed consent for participation in observational study (incl. telephone follow-ups)
* Not simultaneously participating in any randomized trial
* At least one ECG-documented, symptomatic, typical atrial flut-ter episode >30sec.
* Isthmus ablation conducted in association with other ablation procedures (e.g. for atrial fibrillation) is permitted

Exclusion Criteria:

* Any prior AFL ablation
* Acute reversible causes for atrial flutter (e.g. acute myocarditis)
* Tricuspid valve replacement
* Right atrial thrombus
* Present pregnancy or breastfeeding woman
* Drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with acute atrial flutter (AFL) and indication for AFL ablation
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Cumulative time [seconds] of radiofrequency catheter ablation and energy [Joule] delivery to achieve bidirectional isthmus block | 1 day
  evaluate radiofrequency catheter ablation of atrial flutter, i.e. the combination of MVG ablation strategy and the IntellaTip Mifi XP 8 mm sensor technology in right atrial ablation in patients with atrial flutterbidirectional isthmus block

SECONDARY OUTCOMES:
Safety | 6 months
  Number of patients with cardiovascular and cerebrovascular events
Effectiveness | 6 months
  Number of patients with recurrence of atrial flutter and/or re-ablation of atrial flutter

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Lewalter, MD, PhD, Principal Investigator — Head, Dept. of Medicine-Cardiology and Intensive Care

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish data in scientific journal